CLINICAL TRIAL: NCT06624033
Title: Single-blind, Randomized, Cross-over Comparative Bioavailability Study About the Kinetics of Plasma Amino Acid Concentrations Subsequent to the Consumption of Innovative Legume-based Products.
Brief Title: Bioavailability of Legume Proteins in Differents Products
Acronym: LEG'UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Principal Investigator, Adeline BLOT, Clinical Research Associate, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CRNH 1 -2020
Record Dates: First submitted 2020-11-09; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Men
Keywords: amino acid; legume; pea; protein
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: participants may receive 6 products in 6 interventions sequentially during the protocol
Who Masked: Participant
Masking Description: single-centre randomized, cross-over controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Chocolate cake with peas (Experimental): the subjects will consume the test meals (arm title)
  Interventions: Other: amino acids kinetics
- Biscuit with peas (Experimental): the subjects will consume the test meals (arm title).
  Interventions: Other: amino acids kinetics
- chopped steack with peas (Experimental): the subjects will consume the test meals (arm title).
  Interventions: Other: amino acids kinetics
- Chocolate cake with gluten (Placebo Comparator): the subjects will consume the test meals (arm title)
  Interventions: Other: amino acids kinetics
- biscuit with gluten (Placebo Comparator): the subjects will consume the test meals (arm title).
  Interventions: Other: amino acids kinetics
- chopped steack (Placebo Comparator): the subjects will consume the test meals (arm title).
  Interventions: Other: amino acids kinetics

INTERVENTIONS:
Other: amino acids kinetics — After a fasting blood sample (T0), the subjects will consume one of the test meals. Nine samples will be then collected at several times after meal ingestion.
  On these samples, plasma concentrations of amino acids, insulin, blood sugar, lipid balance and inflammatory markers will be measured.

SUMMARY:
The use of pea proteins could be interesting in specific foods. Indeed, these proteins could have great nutritional quality, with good amino acid profile. Therefore, the investigators study the bioavailability of protein and post-prandial variation of metabolic markers following consumption of pea protein-enriched products in healthy young subjects.

Main Objective is to compare plasma kinetics of leucine.

DETAILED DESCRIPTION:
The written agreement of the subjects will be obtained after information on the aims, nature and possible risks of the study.

Before inclusion, the volunteers will be subjected to a medical check-up at the Nutritional Exploration Unit which includes an examination of personal and family history and current drug treatments, as well as a standard medical examination and a blood test for a biological check-up. Compliance with the inclusion/ exclusion criteria will be verified during this review.

Volunteers included in the protocol will go to the Clinical Pharmacology Center (CPC) to perform the tests. At each visit, each volunteer will receive one of the six products.

The volunteer will be reviewed six times for the realization of a kinetics. First, three visits will be made with at least 7 days apart (wash out period). Then, after a 15-day break, three others visits will be organized spaced at least 7 days apart. The day before each visit, the evening meal will be standardized and eaten before 9 pm. A short catheter will be placed in a vein in the forearm for blood samples. After a fasting blood sample (T0), the subjects will consume one of the test meals. Nine samples will be then collected at several times after meal ingestion.

On these samples, plasma concentrations of amino acids, insulin, blood sugar, lipid balance and inflammatory markers will be measured. Any intercurrent events will be noted in the observation book. The test meal sequence will be randomly assigned to subjects (generating a random list) prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Major male volunteers under 30 (<30)
* Body mass index between 22 and 28 kg/m²
* Subjects considered healthy by investigator based on the examination, medical and clinical examination,
* biological check up considered compatible with study participation
* person who is in the position to sign informed consent

Exclusion Criteria:

* Subject with a particular diet (vegetarians, vegans, nutritional supplements, etc.),
* Subject weight < 60 kg
* Subject refusing to consume one of the proposed products or the test meal
* Subject with a food allergy(s) to one or more components of the study products (gluten, legumes, etc.), or with a contribution to the consumption of these products.
* Subject with tumor pathology, inflammatory, moderate to severe kidney failure, malabsorption syndrome,
* Subject being under drug treatment or dietary supplement that may influence the results of kinetics: treatments that may affect gastric emptying, intestinal absorption (smectite-based intestinal dressings, etc.), insulin and blood sugar, Oral nutritional supplements (NOC), proton pump inhibitors (PPIs), corticosteroids, nonsteroidal anti-inflammatory drugs, antibiotics for less than a month,
* Subject with diabetes or dyslipidemia,
* Subject with a heavy medical or surgical history that may pose a risk to the volunteer under the protocol,
* Subject who has undergone surgery that may interfere with the objectives of the study (at the discretion of the investigating physician) within 3 months preceding the study,
* Person refusing to be registered on the National File of Healthy Volunteers of the Ministry of Health,
* Major subject under trusteeship or with limited rights,
* Subject not affiliated with social security,
* Subject during the exclusion period of a previous study (after verification in the Biomedical Research Volunteers File).

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Changes in the plasma concentrations of leucinemia | 0 minute before the consumption of the test meals
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point before (basal)
Changes in the plasma concentrations of leucinemia | 15 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 15 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 30 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 30 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 60 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 60 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 90 minutes after ingestion meals
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 90 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 120 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 120 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 150 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 150 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 180 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 180 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 210 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 210 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 240 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 240 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 270 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 270 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 300 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product).One point at 300 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of leucinemia | 360 minutes after ingestion
  Maximum total plasma concentration of leucinemia measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 360 minutes after the consumption of one of the 6 test periods.

SECONDARY OUTCOMES:
Changes in the plasma concentrations of the others amino acids | 0 minute before the consumption of the test meals,
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point before (basal) the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 15 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 15 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 30 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 30 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 45 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 45 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 60 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 60 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 90 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 90 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 120 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 120 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 180 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 180 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 210 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 210 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 240 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 240 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 270 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 270 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 300 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 300 minutes after the consumption of one of the 6 test periods.
Changes in the plasma concentrations of the others amino acids | 360 minutes after ingestion
  Maximum total plasma concentration of amino-acid measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 360 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 0 minute before the consumption of the test meals
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point before (basal) the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 15 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 15 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 30 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 30 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 45 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 45 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 60 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 60 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 90 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 90 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 120 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 120 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 150 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 150 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 180 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 180 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 210 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 210 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 240 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 240 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 270 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 270 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 300 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 300 minutes after the consumption of one of the 6 test periods.
Changes of Blood sugar levels | 360 minutes after ingestion
  Maximum total concentration of blood sugar measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 360 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 0 minute before the consumption of the test meals
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point before (basal) the consumption of one of the 6 test periods.
Changes of insulin levels | 15 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 15 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 30 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 30 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 45 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 45 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 60 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 60 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 90 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 90 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 120 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 120 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 150 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 150 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 180 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 180 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 210 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 210 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 240 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 240 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 270 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 270 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 300 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 300 minutes after the consumption of one of the 6 test periods.
Changes of insulin levels | 360 minutes after ingestion
  Maximum total concentration of insulin measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 360 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 0 minute before the consumption of the test meals
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point before (basal) the consumption of one of the 6 test periods.
Changes lipid profile | 15 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 15 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 30 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 30 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 45 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 45 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 60 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 60 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 90 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 90 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 120 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 120 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 150 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 150 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 180 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 180 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 210 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 210 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 240 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 240 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 270 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 270 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 300 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 300 minutes after the consumption of one of the 6 test periods.
Changes lipid profile | 360 minutes after ingestion
  Maximum total concentration of lipid profile measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 360 minutes after the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 0 minute before the consumption of the test meals
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point before (basal) the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 15 minutes after ingestion
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 15 minutes after the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 30 minutes after ingestion
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 30 minutes after the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 60 minutes after ingestion
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 60 minutes after the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 90 minutes after ingestion
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 90 minutes after the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 120 minutes after ingestion
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 120 minutes after the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 150 minutes after ingestion
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 150 minutes after the consumption of one of the 6 test periods.
Changes of pro-inflammatory cytokines (TNF α, IL-6 and IL-1β) | 240 minutes after ingestion
  Maximum total plasma concentration of of the pro-inflammatory cytokines measured during different points of the 6 hours of the kinetics (one kinetic / type of product). One point at 240 minutes after the consumption of one of the 6 test periods.
Areas under curves | 0 minute before the consumption of the test meals
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 15 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 30 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 60 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 90 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 120 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 180 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 240 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 300 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals
Areas under curves | 360 minutes after ingestion
  maximum concentration and time to reach this concentration will be compared between test meals

CONTACTS AND LOCATIONS:
Overall Officials: Marine Gueugneau, Phd, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre de Recherche en Nutrition Clinique d'Auvergne, Clermont-Ferrand, Auvergne, France